CLINICAL TRIAL: NCT06247020
Title: Metabolic Effects of Oral Sodium Butyrate Supplementation on Overweight Individuals: a Pilot Study
Brief Title: Metabolic Effects of Oral Sodium Butyrate Supplementation on Overweight Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, rivellese angela, Full Professor, Federico II University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 368/19
Record Dates: First submitted 2024-01-15; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Glucose Metabolism Disorders; Overweight or Obesity
Keywords: butyrate; sodium butyrate; short chain fatty acids; glucose; insulin
MeSH Terms: conditions — Glucose Metabolism Disorders; Overweight; Obesity; Insulin Resistance | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral sodium-butyrrate supplementation (Experimental): Participants consumed 8 capsules of sodium butyrate per day for a week. The capsules were consumed with main meals (2 for breakfast, 2 for lunch and 2 for dinner). Each capsule contained 200 mg of sodium butyrate, for a total of 1.6 grams of sodium butyrate per day.
  Interventions: Dietary Supplement: Supplementation with sodium- butyrrate
- Placebo (Placebo Comparator): Participants consumed 8 capsules of placebo. The capsules were consumed with main meals (2 for breakfast, 2 for lunch and 2 for dinner). Each capsule contained cornstarch
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Supplementation with sodium- butyrrate — Oral supplementation with sodium butyrrate capsules
  Arms: Oral sodium-butyrrate supplementation
Dietary Supplement: Placebo — Oral supplementation with placebo capsules
  Arms: Placebo

SUMMARY:
Numerous evidences suggest an important role of short-chain fatty acids, produced by the intestinal fermentation of dietary fibers by the intestinal microbiota, in the modulation of various biological functions relevant to human health. In particular, butyrate, in addition to its trophic action on enterocytes, could improve insulin sensitivity and increase GLP-1 secretion, suggesting a possible role in the modulation of glucose metabolism. However, to date, very few randomized controlled trials (RCTs) have observed a significant increase in plasma butyrate concentrations in humans after nutritional interventions with high-fiber diets or foods. Butyrate occurs naturally in some foods, such as milk and dairy products, where it is often associated with sodium, becoming sodium butyrate. Therefore, recent studies suggest the use of oral sodium butyrate supplements in order to obtain a significant increase in butyrate plasma concentrations able to exert the potential beneficial effects related to them. To date, few studies have investigated the effect of oral sodium butyrate supplementation on glucose metabolism in healthy or overweight individuals, individuals at high cardiometabolic risk, and individuals with type 2 diabetes. Therefore, the purpose of this pilot study is to evaluate the effects of oral sodium butyrate supplementation, versus placebo, on glucose tolerance and insulin sensitivity in a group of overweight/obese individuals and the mechanisms underlying these effects.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index: 25-30 kg/m2

Exclusion Criteria:

* type 2 diabetes,
* treatment with antibiotics within the past 3 months
* history of gastrointestinal diseases (Inflammatory bowel disease, Crohn's disease, malabsorption etc )
* cardiovascular events (myocardial infarction or stroke) during the 6-12 months prior to the study
* thyroid disorders not controlled by drug therapy,
* kidney (creatinine >1.7 mg/dl or proteinuria) and liver diseases (ALT/AST >twice the upper limits)
* anaemia (Hb <12 g /dl)
* pregnancy or breastfeeding,
* celiac disease, cancer or any other chronic disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Plasma glucose | one week
  The primary outcome of the study is the improvement of the glucose response during an oral glucose tolerance test (OGTT) after the supplementation with sodium butyrate, without changes in body weight

SECONDARY OUTCOMES:
Plasma insulin | one week
  The secondary outcome of the study is the improvement of the insulin response during an oral glucose tolerance test (OGTT) after the supplementation with sodium butyrate, without changes in body weightglycemic and insulinemic response during an OGTT separately in men and women

CONTACTS AND LOCATIONS:
Overall Officials: Angela Albarosa Rivellese, PO, Principal Investigator — Federico II University
Locations (1):
- Federico II University, Department of Clinical Medicine and Surgery, Naples, Italy